CLINICAL TRIAL: NCT05127304
Title: Health Care Resource Utilization, Cost and Other Outcomes of Patients Diagnosed With COPD Initiating Tiotropium Bromide/Olodaterol Versus Fluticasone Furoate/Umeclidinium/Vilanterol
Brief Title: A Study Using US Medical and Pharmacy Claim Records to Compare the Resource Use, Cost, and Outcomes of People With COPD Who Take Either Tiotropium + Olodaterol or Fluticasone + Umeclidinium + Vilanterol
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1237-0113
Record Dates: First submitted 2021-11-12; First posted 2021-11-19 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; olodaterol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Tiotropium bromide/Olodaterol (TIO/OLO): Chronic Obstructive Pulmonary Disease (COPD) patients with ≥30 consecutive days with TIO/OLO initiated during the patient identification period of 01 June 2015 to 30 November 2019 and ≥40 years of age as of the year of the index date. The index date was the date of the TIO/OLO pharmacy claim that started the ≥30 consecutive days with the medication.
  Interventions: Device: Stiolto Respimat; Drug: Tiotropium Bromide/Olodaterol
- Fluticasone furoate/Umeclidinium/Vilanterol (FF/UMEC/VI): Chronic Obstructive Pulmonary Disease (COPD) patients with ≥30 consecutive days with FF/UMEC/VI initiated during the patient identification period of 01 June 2015 to 30 November 2019 and ≥40 years of age as of the year of the index date. The index date was the date of the FF/UMEC/VI pharmacy claim that started the ≥30 consecutive days with the medication.
  Interventions: Device: Trelegy Ellipta; Drug: Furoate/Umeclidinium/Vilanterol

INTERVENTIONS:
Device: Trelegy Ellipta — Trelegy Ellipta with Furoate/Umeclidinium/Vilanterol
  Groups: Fluticasone furoate/Umeclidinium/Vilanterol (FF/UMEC/VI)
Device: Stiolto Respimat — Stiolto Respimat with Tiotropium Bromide/Olodaterol
  Groups: Tiotropium bromide/Olodaterol (TIO/OLO)
Drug: Furoate/Umeclidinium/Vilanterol — Furoate/Umeclidinium/Vilanterol
  Groups: Fluticasone furoate/Umeclidinium/Vilanterol (FF/UMEC/VI)
Drug: Tiotropium Bromide/Olodaterol — Tiotropium Bromide/Olodaterol
  Groups: Tiotropium bromide/Olodaterol (TIO/OLO)

SUMMARY:
The purpose of this study is to estimate disease-related and all-cause burden and clinical outcomes of interest following initiation of chronic obstructive lung disease (COPD) maintenance therapy with Tiotropium Bromide/Olodaterol (TIO/OLO) or Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI).

ELIGIBILITY:
Inclusion Criteria:

* ≥30 consecutive days with Tiotropium Bromide/Olodaterol (TIO/OLO) or Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI) initiated during the patient identification period of 01 June 2015 to 30 November 2019. The index date will be the date of the TIO/OLO or FF/UMEC/VI pharmacy claim that starts the ≥30 consecutive days with the medication.
* >1 facility claim with a diagnosis of chronic obstructive lung disease (COPD) in the primary position or ≥2 professional claims with a diagnosis code for COPD in any position on separate dates of service during the study period
* ≥40 years of age as of the year of the index date
* Continuous enrollment with medical and pharmacy coverage for 12 months prior to and including the index date (baseline period)
* Continuous enrollment with medical and pharmacy coverage for ≥30 days following the index date and without discontinuation of the index medication or switch to a non-index regimen (follow-up period); discontinuation and switch as defined in the protocol.

Exclusion Criteria:

* ≥2 medical claims with a diagnosis code for asthma, cystic fibrosis, lung cancer, or interstitial lung disease in any position on separate dates of service during the baseline period
* Pharmacy claims for both TIO/OLO and FF/UMEC/VI on the index date
* A pharmacy claim for any non-index COPD maintenance medication on the index date, defined as: long-acting muscarinic antagonists (LAMA) monotherapy; long-acting beta2 agonists (LABA) monotherapy; inhaled corticosteroids (ICS) monotherapy; fixed-dose combination (FDC) ICS/LABA, or FDC LAMA/LABA
* Free or fixed dose LAMA+LABA maintenance therapy defined as ≥7 consecutive days of overlapping days' supply with a LAMA and LABA during a 6-month pre-index period, excluding the index date

  -- Flags will be created to identify patients excluded for baseline LAMA/LABA use overall and specifically for each FDC LAMA/LABA medication
* Free or fixed dose triple therapy (TT) defined as ≥7 consecutive days of overlapping days' supply with an ICS, LABA, and LAMA during a 6-month pre-index period, excluding the index date
* ≥1 medical claim with a procedure code for lung volume reduction during the study period
* Unknown age, gender, or business line, or unknown/other geographic region

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample will include commercial and Medicare Advantage Part D (MAPD) health plan members diagnosed with COPD
Sampling Method: Non-Probability Sample
Enrollment: 11316 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-02-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Optum, Eden Prairie, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Sethi S, Palli SR, Bengtson LGS, Buysman EK, Clark B, Sargent A, Shaikh A, Ferguson GT. Clinical and economic outcomes in patients with chronic obstructive pulmonary disease initiating maintenance therapy with tiotropium bromide/olodaterol or fluticasone furoate/umeclidinium/vilanterol. J Manag Care Spec Pharm. 2023 Jul;29(7):791-806. doi: 10.18553/jmcp.2023.22373. Epub 2023 May 3. PMID 37133429
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a non-interventional study using existing data from commercial and Medicare Advantage Part D (MAPD) beneficiaries, using administrative claims data for the period of 01 June 2015 through 30 November 2019.
Pre-assignment Details: Only subjects that met all inclusion and none of the exclusion criteria were included.
Period: Overall Study
Arm/Group | Tiotropium Bromide/Olodaterol (TIO/OLO) | Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI)
Started (Overall post matched) | 5658 | 5658
Completed | 5658 | 5658
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Matched Overall Population: Stratified propensity score matching (PSM), using an exact match on some variables and a propensity score match on the others, was used to control for possible confounding of the association between the outcomes and treatment with TIO/OLO or FF/UMEC/VI. Patients were matched in a 1:1 ratio of TIO/OLO to FF/UMEC/VI.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tiotropium Bromide/Olodaterol (TIO/OLO) | Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI) | Total
Number analyzed (Participants) | 5658 | 5658 | 11316
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.69 (8.69) | 71.75 (8.61) | 71.72 (8.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2846 | 2866 | 5712
  Male | 2812 | 2792 | 5604
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 311 | 281 | 592
  Non- Hispanic Black | 731 | 740 | 1471
  Non- Hispanic White | 4015 | 3815 | 7830
  Non- Hispanic Asian | 78 | 62 | 140
  Other/unknown | 523 | 760 | 1283

OUTCOME MEASURES:

1. Primary Outcome: All-cause Health Care Resource Utilization
Description: All-cause health care resource utilization. Annualized population averages of visits for each of the following categories is reported:
  * Ambulatory visits
  * Office visits
  * Outpatient visits
  * Emergency room visits
  * Inpatient visits
  * Other medical visits (included services like independent laboratory, home health, durable medical equipment, etc.) Annualized population averages of visits were calculated as: ([sum of all visits for all individuals during the follow-up period] / [sum of follow-up on-treatment time in years (365 days) for all individuals]).
Time Frame: Follow-up period (started on the day after the index date, with a minimum of 30-days duration (index date + 1 through index date+30) up to a maximum of 12 months duration (index date + 1 through index date +365).
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: visits/year
Arm/Group | Tiotropium Bromide/Olodaterol (TIO/OLO) | Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI)
Number analyzed (Participants) | 5658 | 5658
visits/year
  Ambulatory visits | 32.54 [31.44 to 33.64] | 32.91 [31.84 to 33.97]
  Office visits | 17.80 [17.25 to 18.35] | 17.57 [17.08 to 18.06]
  Outpatient visits | 14.82 [13.95 to 15.69] | 15.42 [14.55 to 16.28]
  Emergency room visits | 1.26 [1.17 to 1.35] | 1.39 [1.29 to 1.50]
  Inpatient visits | 0.45 [0.41 to 0.48] | 0.48 [0.44 to 0.52]
  Other medical visits | 10.09 [9.69 to 10.49] | 10.48 [10.07 to 10.89]
Statistical Analysis 1: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Ambulatory visits; Test type: Other; p = 0.639, Weighted clustered linear regression
Statistical Analysis 2: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Office visits; Test type: Other; p = 0.535, Weighted clustered linear regression
Statistical Analysis 3: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Outpatient visits; Test type: Other; p = 0.337, Weighted clustered linear regression
Statistical Analysis 4: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Emergency room visits; Test type: Other; p = 0.058, Weighted clustered linear regression
Statistical Analysis 5: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Inpatient visits; Test type: Other; p = 0.192, Weighted clustered linear regression
Statistical Analysis 6: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Other medical visits; Test type: Other; p = 0.176, Weighted clustered linear regression

2. Primary Outcome: All-cause Health Care Resource Utilization: Inpatient Days
Description: All-cause health care resource utilization: Inpatient days. Annualized population averages of inpatient days is reported.
  Annualized population averages of inpatient days were calculated as: ([sum of all inpatient days for all individuals during the follow-up period] / [sum of follow-up on-treatment time in years (365 days) for all individuals]).
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: inpatient days/year
Arm/Group | Tiotropium Bromide/Olodaterol (TIO/OLO) | Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI)
Number analyzed (Participants) | 5658 | 5658
inpatient days/year | 4.30 [3.80 to 4.79] | 4.68 [4.12 to 5.24]
Statistical Analysis 1: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Test type: Other; p = 0.313, Weighted clustered linear regression

3. Primary Outcome: All-cause Health Care Resource Utilization: Pharmacy Fills
Description: All-cause health care resource utilization: Pharmacy fills. Annualized population averages for pharmacy fills is reported.
  Annualized population averages of pharmacy fills were calculated as:([sum of all pharmacy fills for all individuals during the follow-up period] / [sum of follow-up on-treatment time in years (365 days) for all individuals]).
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: pharmacy fills/year
Arm/Group | Tiotropium Bromide/Olodaterol (TIO/OLO) | Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI)
Number analyzed (Participants) | 5658 | 5658
pharmacy fills/year | 59.39 [58.05 to 60.73] | 57.13 [55.75 to 58.52]
Statistical Analysis 1: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Test type: Other; p = 0.021, Weighted clustered linear regression

4. Primary Outcome: COPD-related Health Care Resource Utilization
Description: Chronic Obstructive Pulmonary Disease (COPD)-related (medical claims with a diagnosis for COPD in any position and pharmacy claims for a COPD-related treatment, including COPD-guideline recommended antibiotics) health care resource utilization. Population annualized averages of visits for each of the following categories is reported:
  * Ambulatory visits
  * Office visits
  * Outpatient visits
  * Emergency room visits
  * Inpatient visits
  * Other medical visits (included services like independent laboratory, home health, durable medical equipment, etc.).
  Annualized population averages of visits were calculated as: ([sum of all visits for all individuals during the follow-up period] / [sum of follow-up on-treatment time in years (365 days) for all individuals]).
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: visits/year
Arm/Group | Tiotropium Bromide/Olodaterol (TIO/OLO) | Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI)
Number analyzed (Participants) | 5658 | 5658
visits/year
  Ambulatory visits | 8.77 [8.30 to 9.23] | 9.56 [9.05 to 10.08]
  Office visits | 3.92 [3.80 to 4.05] | 4.07 [3.93 to 4.20]
  Outpatient visits | 4.85 [4.42 to 5.28] | 5.51 [5.03 to 5.98]
  Emergency room visits | 0.65 [0.59 to 0.71] | 0.65 [0.59 to 0.71]
  Inpatient visits | 0.39 [0.36 to 0.42] | 0.44 [0.41 to 0.48]
  Other medical visits | 4.28 [4.04 to 4.53] | 4.87 [4.61 to 5.13]
Statistical Analysis 1: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Ambulatory visits; Test type: Other; p = 0.022, Weighted clustered linear regression
Statistical Analysis 2: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Office visits; Test type: Other; p = 0.124, Weighted clustered linear regression
Statistical Analysis 3: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Outpatient visits; Test type: Other; p = 0.043, Weighted clustered linear regression
Statistical Analysis 4: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Emergency room visits; Test type: Other; p = 0.990, Weighted clustered linear regression
Statistical Analysis 5: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Inpatient visits; Test type: Other; p = 0.039, Weighted clustered linear regression
Statistical Analysis 6: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Other medical visits; Test type: Other; p < 0.001, Weighted clustered linear regression

5. Primary Outcome: COPD-related Health Care Resource Utilization: Inpatient Days
Description: Chronic Obstructive Pulmonary Disease (COPD)-related (medical claims with a diagnosis for COPD in any position and pharmacy claims for a COPD-related treatment, including COPD-guideline recommended antibiotics) health care resource utilization: Inpatient days. Population annualized averages of inpatient days is reported.
  Annualized population averages of inpatient days were calculated as: ([sum of all inpatient days for all individuals during the follow-up period] / [sum of follow-up on-treatment time in years (365 days) for all individuals]).
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: inpatient days/year
Arm/Group | Tiotropium Bromide/Olodaterol (TIO/OLO) | Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI)
Number analyzed (Participants) | 5658 | 5658
inpatient days/year | 3.91 [3.43 to 4.38] | 4.42 [3.87 to 4.97]
Statistical Analysis 1: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Test type: Other; p = 0.163, Weighted clustered linear regression

6. Primary Outcome: COPD-related Health Care Resource Utilization: Pharmacy Fills
Description: Chronic Obstructive Pulmonary Disease (COPD)-related (medical claims with a diagnosis for COPD in any position and pharmacy claims for a COPD-related treatment, including COPD-guideline recommended antibiotics) health care resource utilization. Population annualized averages for pharmacy fills is reported.
  Annualized population averages of pharmacy fills were calculated as: ([sum of all pharmacy fills for all individuals during the follow-up period] / [sum of follow-up on-treatment time in years (365 days) for all individuals]).
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: pharmacy fills/year
Arm/Group | Tiotropium Bromide/Olodaterol (TIO/OLO) | Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI)
Number analyzed (Participants) | 5658 | 5658
pharmacy fills/year | 15.48 [15.20 to 15.77] | 15.08 [14.82 to 15.35]
Statistical Analysis 1: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Test type: Other; p = 0.037, Weighted clustered linear regression

7. Primary Outcome: COPD and/or Pneumonia-related Health Care Resource Utilization
Description: Chronic Obstructive Pulmonary Disease (COPD) and/or pneumonia-related health care resource utilization (medical claims with a diagnosis for COPD, pneumonia, or acute bronchitis/bronchiolitis in any position and pharmacy claims for a COPD-related treatment, including COPD-guideline recommended antibiotics).
  Population annualized averages of visits in each of the following categories is reported:
  * Ambulatory visits
  * Office visits
  * Outpatient visits
  * Emergency room visits
  * Inpatient visits
  * Other medical visits (independent laboratory, home health, durable medical equipment, etc.)
  Population annualized averages of visits were calculated as: ([sum of all visits for all individuals during the follow-up period] / [sum of follow-up on-treatment time in years (365 days) for all individuals]).
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: visits/year
Arm/Group | Tiotropium Bromide/Olodaterol (TIO/OLO) | Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI)
Number analyzed (Participants) | 5658 | 5658
visits/year
  Ambulatory visits | 9.01 [8.54 to 9.48] | 9.85 [9.33 to 10.37]
  Office visits | 4.04 [3.91 to 4.16] | 4.19 [4.06 to 4.33]
  Outpatient visits | 4.98 [4.55 to 5.42] | 5.67 [5.19 to 6.15]
  Emergency room visits | 0.70 [0.63 to 0.76] | 0.70 [0.64 to 0.76]
  Inpatient visits | 0.40 [0.37 to 0.43] | 0.45 [0.42 to 0.49]
  Other medical visits | 4.36 [4.11 to 4.61] | 4.94 [4.68 to 5.20]
Statistical Analysis 1: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Ambulatory visits; Test type: Other; p = 0.017, Weighted clustered linear regression
Statistical Analysis 2: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Office visits; Test type: Other; p = 0.098, Weighted clustered linear regression
Statistical Analysis 3: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Outpatient visits; Test type: Other; p = 0.036, Weighted clustered linear regression
Statistical Analysis 4: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Emergency room visits; Test type: Other; p = 0.894, Weighted clustered linear regression
Statistical Analysis 5: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Inpatient visits; Test type: Other; p = 0.036, Weighted clustered linear regression
Statistical Analysis 6: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Other medical visits; Test type: Other; p = 0.001, Weighted clustered linear regression

8. Primary Outcome: COPD and/or Pneumonia-related Health Care Resource Utilization: Inpatient Days
Description: Chronic Obstructive Pulmonary Disease (COPD) and/or pneumonia-related health care resource utilization (medical claims with a diagnosis for COPD, pneumonia, or acute bronchitis/bronchiolitis in any position and pharmacy claims for a COPD-related treatment, including COPD-guideline recommended antibiotics).
  Population annualized averages of inpatient days is reported.
  Population annualized averages of inpatient days were calculated as: ([sum of all inpatient days for all individuals during the follow-up period] / [sum of follow-up on-treatment time in years (365 days) for all individuals]).
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: inpatient days/year
Arm/Group | Tiotropium Bromide/Olodaterol (TIO/OLO) | Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI)
Number analyzed (Participants) | 5658 | 5658
inpatient days/year | 3.97 [3.49 to 4.45] | 4.49 [3.94 to 5.05]
Statistical Analysis 1: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Test type: Other; p = 0.162, Weighted clustered linear regression

9. Primary Outcome: COPD and/or Pneumonia-related Health Care Resource Utilization: Pharmacy Fills
Description: Chronic Obstructive Pulmonary Disease (COPD) and/or pneumonia-related health care resource utilization (medical claims with a diagnosis for COPD, pneumonia, or acute bronchitis/bronchiolitis in any position and pharmacy claims for a COPD-related treatment, including COPD-guideline recommended antibiotics).
  Population annualized averages of pharmacy fills is reported.
  Population annualized averages of pharmacy fills were calculated as: ([sum of all pharmacy fills for all individuals during the follow-up period] / [sum of follow-up on-treatment time in years (365 days) for all individuals]).
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: pharmacy fills/year
Arm/Group | Tiotropium Bromide/Olodaterol (TIO/OLO) | Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI)
Number analyzed (Participants) | 5658 | 5658
pharmacy fills/year | 15.48 [15.20 to 15.77] | 15.08 [14.82 to 15.35]
Statistical Analysis 1: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Test type: Other; p = 0.037, Weighted clustered linear regression

10. Primary Outcome: Pneumonia-related Health Care Resource Utilization
Description: Pneumonia-related health care resource utilization: This utilization was calculated for medical claims with a diagnosis for pneumonia in any position.
  Population annualized averages of visits in each of the following categories is reported:
  * Ambulatory visits
  * Office visits
  * Outpatient visits
  * Emergency room visits
  * Inpatient visits
  * Other medical visits (independent laboratory, home health, durable medical equipment, etc.)
  Population annualized averages of visits were calculated as: ([sum of all visits for all individuals during the follow-up period] / [sum of follow-up on-treatment time in years (365 days) for all individuals]).
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: visits/year
Arm/Group | Tiotropium Bromide/Olodaterol (TIO/OLO) | Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI)
Number analyzed (Participants) | 5658 | 5658
visits/year
  Ambulatory visits | 0.49 [0.38 to 0.59] | 0.66 [0.51 to 0.81]
  Office visits | 0.13 [0.10 to 0.15] | 0.15 [0.13 to 0.18]
  Outpatient visits | 0.36 [0.26 to 0.46] | 0.50 [0.37 to 0.64]
  Emergency room visits | 0.10 [0.08 to 0.11] | 0.11 [0.09 to 0.13]
  Inpatient visits | 0.12 [0.10 to 0.13] | 0.15 [0.13 to 0.17]
  Other medical visits | 0.12 [0.07 to 0.16] | 0.12 [0.09 to 0.16]
Statistical Analysis 1: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Ambulatory visits; Test type: Other; p = 0.065, Weighted clustered linear regression
Statistical Analysis 2: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Office visits; Test type: Other; p = 0.102, Weighted clustered linear regression
Statistical Analysis 3: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Outpatient visits; Test type: Other; p = 0.100, Weighted clustered linear regression
Statistical Analysis 4: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Emergency room visits; Test type: Other; p = 0.189, Weighted clustered linear regression
Statistical Analysis 5: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Inpatient visits; Test type: Other; p = 0.024, Weighted clustered linear regression
Statistical Analysis 6: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Other medical visits; Test type: Other; p = 0.767, Weighted clustered linear regression

11. Primary Outcome: Pneumonia-related Health Care Resource Utilization: Inpatient Days
Description: Pneumonia-related health care resource utilization: This utilization was calculated for medical claims with a diagnosis for pneumonia in any position.
  Population annualized averages of inpatient days is reported.
  Population annualized averages of inpatient days were calculated as: ([sum of all inpatient days for all individuals during the follow-up period] / [sum of follow-up on-treatment time in years (365 days) for all individuals]).
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: inpatient days/year
Arm/Group | Tiotropium Bromide/Olodaterol (TIO/OLO) | Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI)
Number analyzed (Participants) | 5658 | 5658
inpatient days/year | 1.72 [1.36 to 2.08] | 1.98 [1.56 to 2.40]
Statistical Analysis 1: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Test type: Other; p = 0.357, Weighted clustered linear regression

12. Primary Outcome: COPD or Pneumonia-attributable Health Care Resource Utilization
Description: COPD or pneumonia-attributable health care resource utilization: This utilization was calculated for medical claims with a diagnosis for COPD, pneumonia, or acute bronchitis/bronchiolitis in the primary position or a diagnosis for acute respiratory failure in the primary position and a diagnosis for COPD, pneumonia, or acute bronchitis/bronchiolitis in a non-primary position and pharmacy claims for a COPD-related treatment, including COPD-guideline recommended antibiotics.
  Population annualized averages of visits in each of the following categories is reported:
  * Ambulatory visits
  * Office visits
  * Outpatient visits
  * Emergency room visits
  * Inpatient visits
  * Other medical visits (independent laboratory, home health, durable medical equipment, etc.)
  Population annualized averages of visits were calculated as: ([sum of all visits for all individuals during the follow-up period] / [sum of follow-up on-treatment time in years (365 days) for all individuals]).
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: visits/year
Arm/Group | Tiotropium Bromide/Olodaterol (TIO/OLO) | Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI)
Number analyzed (Participants) | 5658 | 5658
visits/year
  Ambulatory visits | 4.20 [3.94 to 4.46] | 4.90 [4.55 to 5.25]
  Office visits | 2.09 [2.00 to 2.17] | 2.14 [2.05 to 2.23]
  Outpatient visits | 2.12 [1.88 to 2.35] | 2.77 [2.44 to 3.10]
  Emergency room visits | 0.29 [0.25 to 0.32] | 0.26 [0.23 to 0.30]
  Inpatient visits | 0.24 [0.21 to 0.26] | 0.25 [0.23 to 0.28]
  Other medical visits | 3.82 [3.58 to 4.05] | 4.27 [4.03 to 4.51]
Statistical Analysis 1: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Ambulatory visits; Test type: Other; p = 0.002, Weighted clustered linear regression
Statistical Analysis 2: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Office visits; Test type: Other; p = 0.420, Weighted clustered linear regression
Statistical Analysis 3: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Outpatient visits; Test type: Other; p = 0.002, Weighted clustered linear regression
Statistical Analysis 4: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Emergency room visits; Test type: Other; p = 0.304, Weighted clustered linear regression
Statistical Analysis 5: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Inpatient visits; Test type: Other; p = 0.326, Weighted clustered linear regression
Statistical Analysis 6: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Other medical visits; Test type: Other; p = 0.007, Weighted clustered linear regression

13. Primary Outcome: COPD or Pneumonia-attributable Health Care Resource Utilization: Inpatient Days
Description: COPD or pneumonia-attributable health care resource utilization: This utilization was calculated for medical claims with a diagnosis for COPD, pneumonia, or acute bronchitis/bronchiolitis in the primary position or a diagnosis for acute respiratory failure in the primary position and a diagnosis for COPD, pneumonia, or acute bronchitis/bronchiolitis in a non-primary position and pharmacy claims for a COPD-related treatment, including COPD-guideline recommended antibiotics.
  Population annualized averages of inpatient days is reported.
  Population annualized averages of inpatient days were calculated as: ([sum of all inpatient days for all individuals during the follow-up period] / [sum of follow-up on-treatment time in years (365 days) for all individuals]).
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: inpatient days/year
Arm/Group | Tiotropium Bromide/Olodaterol (TIO/OLO) | Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI)
Number analyzed (Participants) | 5658 | 5658
inpatient days/year | 2.87 [2.43 to 3.31] | 3.08 [2.59 to 3.58]
Statistical Analysis 1: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Test type: Other; p = 0.520, Weighted clustered linear regression

14. Primary Outcome: COPD or Pneumonia-attributable Health Care Resource Utilization: Pharmacy Fills
Description: COPD or pneumonia-attributable health care resource utilization: This utilization was calculated for medical claims with a diagnosis for COPD, pneumonia, or acute bronchitis/bronchiolitis in the primary position or a diagnosis for acute respiratory failure in the primary position and a diagnosis for COPD, pneumonia, or acute bronchitis/bronchiolitis in a non-primary position and pharmacy claims for a COPD-related treatment, including COPD-guideline recommended antibiotics.
  Annualized population averages for pharmacy claims are calculated as the ([sum of all pharmacy fills for all individuals during the follow-up period] / [sum of follow-up on-treatment time in years (365 days) for all individuals]). Wald 95% confidence limits for this ratio used the Taylor expansion to estimate the standard error.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: pharmacy fills/year
Arm/Group | Tiotropium Bromide/Olodaterol (TIO/OLO) | Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI)
Number analyzed (Participants) | 5658 | 5658
pharmacy fills/year | 15.48 [15.20 to 15.77] | 15.08 [14.82 to 15.35]
Statistical Analysis 1: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Test type: Other; p = 0.037, Weighted clustered linear regression

15. Primary Outcome: All-cause Health Care Costs (Insurer + Patient Paid Amounts)
Description: All-cause health care costs were computed from the payer and patient perspective together.
  Annualized population averages of all-cause health care costs in each of the following categories is reported:
  * Medical costs (includes physician office costs, hospital outpatient costs, emergency services costs, inpatient costs, and other costs)
  * Ambulatory
  * Office visits
  * Outpatient visits
  * Emergency room visits
  * Inpatient stay
  * Other medical costs
  * Pharmacy costs
  * Total (medical + pharmacy) costs. Annualized population averages of costs were calculated as: ([sum of all costs for all individuals during the follow-up period] / [sum of follow-up on-treatment time in years (365 days) for all individuals]).
  Costs were adjusted to 2020 dollars using the most recent year of the medical care component of the Consumer Price Index (CPI) to reflect inflation between the date of the claim and 2020.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: dollars/year
Arm/Group | Tiotropium Bromide/Olodaterol (TIO/OLO) | Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI)
Number analyzed (Participants) | 5658 | 5658
dollars/year
  Medical costs | 16911.48 [15847.98 to 17974.99] | 18471.61 [17239.50 to 19703.71]
  Ambulatory costs | 7321.14 [6778.92 to 7863.36] | 7858.06 [7294.85 to 8421.27]
  Office visits costs | 2986.46 [2689.18 to 3283.74] | 3030.56 [2747.15 to 3313.97]
  Outpatient visits costs | 4334.68 [3904.48 to 4764.88] | 4827.50 [4373.94 to 5281.07]
  Emergency room visits costs | 991.35 [905.13 to 1077.57] | 1086.48 [985.78 to 1187.18]
  Inpatient stay costs | 7480.17 [6676.49 to 8283.85] | 8139.51 [7219.72 to 9059.31]
  Other medical costs | 1118.83 [1030.70 to 1206.95] | 1387.55 [1127.10 to 1648.01]
  Pharmacy costs | 10192.10 [9694.69 to 10689.50] | 11963.02 [11348.38 to 12577.66]
  Total (medical + pharmacy) costs | 27103.58 [25871.20 to 28335.96] | 30434.63 [29019.36 to 31849.89]
Statistical Analysis 1: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Medical costs; Test type: Other; p = 0.060, Weighted clustered linear regression
Statistical Analysis 2: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Ambulatory costs; Test type: Other; p = 0.177, Weighted clustered linear regression
Statistical Analysis 3: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Office visits costs; Test type: Other; p = 0.834, Weighted clustered linear regression
Statistical Analysis 4: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Outpatient visits costs; Test type: Other; p = 0.121, Weighted clustered linear regression
Statistical Analysis 5: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Emergency room visits costs; Test type: Other; p = 0.159, Weighted clustered linear regression
Statistical Analysis 6: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Inpatient stay costs; Test type: Other; p = 0.289, Weighted clustered linear regression
Statistical Analysis 7: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Other medical costs; Test type: Other; p = 0.055, Weighted clustered linear regression
Statistical Analysis 8: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Pharmacy costs; Test type: Other; p < 0.001, Weighted clustered linear regression
Statistical Analysis 9: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Total (medical + pharmacy) costs; Test type: Other; p < 0.001, Weighted clustered linear regression

16. Primary Outcome: COPD-related Health Care Costs (Insurer + Patient Paid Amounts)
Description: COPD-related health care costs (HCC) cover the costs for medical claims with a diagnosis for COPD in any position and pharmacy claims for a COPD-related treatment, including COPD-guideline recommended antibiotics. Annualized population averages of COPD-related HCC for the categories below are reported:
  * Medical costs (includes physician office costs, hospital outpatient costs, emergency services costs, inpatient costs, and other costs)
  * Ambulatory
  * Office visits
  * Outpatient visits
  * Emergency room visits
  * Inpatient stay
  * Other medical costs
  * Pharmacy costs
  * Total (medical + pharmacy) costs. Annualized population averages of costs = ([sum of all costs for all individuals during the follow-up period] / [sum of follow-up on-treatment time in years (365 days) for all individuals]).
  Costs are adjusted to 2020 dollars using the most recent year of the medical care component of the Consumer Price Index (CPI) to reflect inflation between the claim date and 2020.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: dollars/year
Arm/Group | Tiotropium Bromide/Olodaterol (TIO/OLO) | Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI)
Number analyzed (Participants) | 5658 | 5658
dollars/year
  Medical costs | 9635.45 [8796.38 to 10474.52] | 10820.05 [9863.73 to 11776.36]
  Ambulatory costs | 2088.43 [1865.20 to 2311.66] | 2278.21 [2098.69 to 2457.72]
  Office visits costs | 468.94 [449.67 to 488.21] | 493.42 [469.73 to 517.12]
  Outpatient visits costs | 1619.49 [1398.51 to 1840.48] | 1784.78 [1608.97 to 1960.60]
  Emergency room visits costs | 426.02 [377.61 to 474.42] | 455.87 [398.69 to 513.05]
  Inpatient stay costs | 6681.35 [5910.54 to 7452.17] | 7596.04 [6700.88 to 8491.21]
  Other medical costs | 439.65 [400.07 to 479.23] | 489.92 [416.29 to 563.56]
  Pharmacy costs | 4729.11 [4675.71 to 4782.50] | 6567.16 [6502.52 to 6631.79]
  Total (medical + pharmacy) costs | 14364.56 [13521.68 to 15207.44] | 17387.20 [16425.26 to 18349.15]
Statistical Analysis 1: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Medical costs; Test type: Other; p = 0.066, Weighted clustered linear regression
Statistical Analysis 2: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Ambulatory costs; Test type: Other; p = 0.193, Weighted clustered linear regression
Statistical Analysis 3: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Office visits costs; Test type: Other; p = 0.117, Weighted clustered linear regression
Statistical Analysis 4: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Outpatient visits costs; Test type: Other; p = 0.250, Weighted clustered linear regression
Statistical Analysis 5: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Emergency room visits costs; Test type: Other; p = 0.431, Weighted clustered linear regression
Statistical Analysis 6: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Inpatient stay costs; Test type: Other; p = 0.129, Weighted clustered linear regression
Statistical Analysis 7: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Other medical costs; Test type: Other; p = 0.236, Weighted clustered linear regression
Statistical Analysis 8: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Pharmacy costs; Test type: Other; p < 0.001, Weighted clustered linear regression
Statistical Analysis 9: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Total (medical + pharmacy) costs; Test type: Other; p < 0.001, Weighted clustered linear regression

17. Primary Outcome: COPD and/or Pneumonia-related Health Care Costs (Insurer + Patient Paid Amounts)
Description: These costs were calculated for medical claims with a diagnosis for COPD, pneumonia, or acute bronchitis/bronchiolitis in any position and pharmacy claims for a COPD-related treatment, including COPD-guideline recommended antibiotics.
  Annualized population averages of costs for categories below is reported:
  * Medical costs (includes physician office costs, hospital outpatient costs, emergency services costs, inpatient costs, and other costs)
  * Ambulatory
  * Office visits
  * Outpatient visits
  * Emergency room visits
  * Inpatient stay
  * Other medical costs
  * Pharmacy costs
  * Total (medical + pharmacy) costs. Annualized population averages=([sum of all costs for all individuals during the follow-up period] / [sum of follow-up on-treatment time in years (365 days) for all individuals]).
  Costs were adjusted to 2020 dollars using the most recent year of the medical care component of the Consumer Price Index (CPI) to reflect inflation between the claim date and 2020.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: dollars/year
Arm/Group | Tiotropium Bromide/Olodaterol (TIO/OLO) | Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI)
Number analyzed (Participants) | 5658 | 5658
dollars/year
  Medical costs | 9828.60 [8983.51 to 10673.68] | 11065.38 [10099.14 to 12031.62]
  Ambulatory costs | 2121.76 [1897.95 to 2345.56] | 2316.77 [2136.31 to 2497.23]
  Office visits costs | 481.16 [461.70 to 500.62] | 508.60 [484.54 to 532.65]
  Outpatient visits costs | 1640.60 [1419.10 to 1862.09] | 1808.18 [1631.62 to 1984.73]
  Emergency room visits costs | 448.83 [399.54 to 498.12] | 482.53 [423.81 to 541.26]
  Inpatient stay costs | 6811.63 [6036.18 to 7587.08] | 7769.37 [6865.53 to 8673.21]
  Other medical costs | 446.38 [406.50 to 486.26] | 496.70 [422.80 to 570.60]
  Pharmacy costs | 4729.11 [4675.71 to 4782.50] | 6567.16 [6502.52 to 6631.79]
  Total (medical + pharmacy) costs | 14557.70 [13708.73 to 15406.67] | 17632.54 [16660.65 to 18604.43]
Statistical Analysis 1: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Medical costs; Test type: Other; p = 0.057, Weighted clustered linear regression
Statistical Analysis 2: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Ambulatory costs; Test type: Other; p = 0.182, Weighted clustered linear regression
Statistical Analysis 3: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Office visits costs; Test type: Other; p = 0.083, Weighted clustered linear regression
Statistical Analysis 4: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Outpatient visits costs; Test type: Other; p = 0.245, Weighted clustered linear regression
Statistical Analysis 5: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Emergency room visits costs; Test type: Other; p = 0.386, Weighted clustered linear regression
Statistical Analysis 6: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Inpatient stay costs; Test type: Other; p = 0.115, Weighted clustered linear regression
Statistical Analysis 7: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Other medical costs; Test type: Other; p = 0.237, Weighted clustered linear regression
Statistical Analysis 8: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Pharmacy costs; Test type: Other; p < 0.001, Weighted clustered linear regression
Statistical Analysis 9: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Total (medical + pharmacy) costs; Test type: Other; p < 0.001, Weighted clustered linear regression

18. Primary Outcome: Pneumonia-related Health Care Costs (Insurer + Patient Paid Amounts)
Description: These costs were calculated for medical claims with a diagnosis for pneumonia in any position.
  Annualized population averages of pneumonia-related health care costs for the categories below is reported:
  * Medical costs (includes physician office costs, hospital outpatient costs, emergency services costs, inpatient costs, and other costs)
  * Ambulatory
  * Office visits
  * Outpatient visits
  * Emergency room visits
  * Inpatient stay
  * Other medical costs
  * Pharmacy costs
  * Total (medical + pharmacy) costs. Annualized population averages=([sum of all costs for all individuals during the follow-up period] / [sum of follow-up on-treatment time in years (365 days) for all individuals]).
  Costs were adjusted to 2020 dollars using the most recent year of the medical care component of the Consumer Price Index (CPI) to reflect inflation between the claim date and 2020.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: dollars/year
Arm/Group | Tiotropium Bromide/Olodaterol (TIO/OLO) | Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI)
Number analyzed (Participants) | 5658 | 5658
dollars/year
  Medical costs | 2857.23 [2293.89 to 3420.58] | 3466.72 [2751.82 to 4181.63]
  Ambulatory costs | 80.62 [55.70 to 105.55] | 98.19 [74.68 to 121.69]
  Office visits costs | 15.03 [11.95 to 18.12] | 18.03 [14.56 to 21.50]
  Outpatient visits costs | 65.59 [42.03 to 89.14] | 80.16 [57.88 to 102.44]
  Emergency room visits costs | 48.91 [34.33 to 63.50] | 51.33 [37.30 to 65.37]
  Inpatient stay costs | 2714.94 [2156.01 to 3273.86] | 3297.65 [2588.62 to 4006.67]
  Other medical costs | 12.77 [3.60 to 21.93] | 19.56 [-1.10 to 40.21]
  Total (medical + pharmacy) costs | 2857.23 [2293.89 to 3420.58] | 3466.72 [2751.82 to 4181.63]
Statistical Analysis 1: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Medical costs; Test type: Other; p = 0.189, Weighted clustered linear regression
Statistical Analysis 2: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Ambulatory costs; Test type: Other; p = 0.314, Weighted clustered linear regression
Statistical Analysis 3: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Office visits costs; Test type: Other; p = 0.203, Weighted clustered linear regression
Statistical Analysis 4: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Outpatient visits costs; Test type: Other; p = 0.379, Weighted clustered linear regression
Statistical Analysis 5: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Emergency room visits costs; Test type: Other; p = 0.815, Weighted clustered linear regression
Statistical Analysis 6: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Inpatient stay costs; Test type: Other; p = 0.205, Weighted clustered linear regression
Statistical Analysis 7: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Other medical costs; Test type: Other; p = 0.556, Weighted clustered linear regression
Statistical Analysis 8: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Total (medical + pharmacy) costs; Test type: Other; p = 0.189, Weighted clustered linear regression

19. Primary Outcome: COPD or Pneumonia-attributable Health Care Costs (Insurer + Patient Paid Amounts)
Description: These costs were calculated for medical claims with a diagnosis for COPD, pneumonia, or acute bronchitis/bronchiolitis in the primary position or a diagnosis for acute respiratory failure in the primary position and a diagnosis for COPD, pneumonia, or acute bronchitis/bronchiolitis in a non-primary position, or pharmacy claims for a COPD-related treatment, including COPD-guideline recommended antibiotics.
  Annualized population averages are reported and were calculated as=([sum of all costs for all individuals during the follow-up period] / [sum of follow-up on-treatment time in years (365 days) for all individuals]).
  Costs were adjusted to 2020 dollars using the most recent year of the medical care component of the Consumer Price Index (CPI) to reflect inflation between the claim date and 2020.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: dollars/year
Arm/Group | Tiotropium Bromide/Olodaterol (TIO/OLO) | Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI)
Number analyzed (Participants) | 5658 | 5658
dollars/year
  Medical costs | 5630.81 [4935.27 to 6326.35] | 6006.47 [5207.40 to 6805.54]
  Ambulatory costs | 517.27 [476.44 to 558.11] | 623.53 [571.43 to 675.62]
  Office visits costs | 231.09 [220.79 to 241.39] | 242.99 [231.84 to 254.15]
  Outpatient visits costs | 286.18 [247.81 to 324.55] | 380.53 [330.93 to 430.14]
  Emergency room visits costs | 153.87 [128.27 to 179.47] | 130.00 [107.47 to 152.53]
  Inpatient stay costs | 4595.72 [3912.28 to 5279.16] | 4885.72 [4099.84 to 5671.61]
  Other medical costs | 363.95 [332.48 to 395.42] | 367.22 [333.81 to 400.62]
  Pharmacy costs | 4729.11 [4675.71 to 4782.50] | 6567.16 [6502.52 to 6631.79]
  Total (medical + pharmacy) costs | 10359.92 [9659.97 to 11059.86] | 12573.62 [11768.74 to 13378.51]
Statistical Analysis 1: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Medical costs; Test type: Other; p = 0.483, Weighted clustered linear regression
Statistical Analysis 2: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Ambulatory costs; Test type: Other; p = 0.002, Weighted clustered linear regression
Statistical Analysis 3: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Office visits costs; Test type: Other; p = 0.123, Weighted clustered linear regression
Statistical Analysis 4: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Outpatient visits costs; Test type: Other; p = 0.003, Weighted clustered linear regression
Statistical Analysis 5: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Emergency room visits costs; Test type: Other; p = 0.170, Weighted clustered linear regression
Statistical Analysis 6: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Inpatient stay costs; Test type: Other; p = 0.582, Weighted clustered linear regression
Statistical Analysis 7: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Other medical costs; Test type: Other; p = 0.887, Weighted clustered linear regression
Statistical Analysis 8: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Pharmacy costs; Test type: Other; p < 0.001, Weighted clustered linear regression
Statistical Analysis 9: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Total (medical + pharmacy) costs; Test type: Other; p < 0.001, Weighted clustered linear regression

20. Primary Outcome: Chronic Obstructive Pulmonary Disease (COPD) Exacerbations
Description: Annualized population averages of COPD exacerbations for the categories below are reported:
  * Any COPD exacerbation
  * Severe COPD exacerbation (defined as an inpatient admission or an emergency room (ER) visit with a COPD diagnosis code in the primary position; or an inpatient admission or an ER visit with a diagnosis code for acute respiratory failure in the primary position and a COPD diagnosis code in any position; or an inpatient admission or an ER visit with a diagnosis code for acute respiratory failure in the primary position + an inpatient admission or an ER visit within ±7 days with a COPD diagnosis code in any position).
  Annualized population averages= ([sum of all exacerbations for all individuals during the follow-up period] / [sum of follow-up on-treatment time in years (365 days) for all individuals]).
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: exacerbations/year
Arm/Group | Tiotropium Bromide/Olodaterol (TIO/OLO) | Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI)
Number analyzed (Participants) | 5658 | 5658
exacerbations/year
  Any COPD exacerbation | 1.02 [0.97 to 1.08] | 0.98 [0.92 to 1.03]
  Severe COPD exacerbation | 0.28 [0.25 to 0.30] | 0.26 [0.24 to 0.29]
Statistical Analysis 1: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Any COPD exacerbation; Test type: Other; p = 0.205, Weighted clustered linear regression
Statistical Analysis 2: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Severe COPD exacerbation; Test type: Other; p = 0.454, Weighted clustered linear regression

21. Secondary Outcome: Percentage of Patients With 30-day All-cause Readmission After COPD Hospitalization
Description: Percentage of patients with 30-day all-cause readmission after Chronic Obstructive Pulmonary Disease (COPD) hospitalization is reported.
  Hospitalizations were classified as COPD-related if they met either of the following 2 criteria:
  * ≥1 diagnosis of COPD in the primary position any time during the acute inpatient stay; or
  * ≥1 diagnosis of acute respiratory failure in the primary position and a diagnosis of acute exacerbation of COPD in a later position on the same claim during an acute inpatient stay.
Time Frame: as for outcome 1
Population: Patients in the Matched Overall Population with a COPD hospitalization during the follow-up period. Matched Overall Population: Stratified propensity score matching (PSM), using an exact match on some variables and a propensity score match on the others, was used to control for possible confounding of the association between the outcomes and treatment with TIO/OLO or FF/UMEC/VI. Patients were matched in a 1:1 ratio of TIO/OLO to FF/UMEC/VI.
Measure: Number; unit: percentage of patients
Arm/Group | Tiotropium Bromide/Olodaterol (TIO/OLO) | Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI)
Number analyzed (Participants) | 191 | 400
percentage of patients | 12.04 | 18.25
Statistical Analysis 1: Comparison: Tiotropium Bromide/Olodaterol (TIO/OLO) vs Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Test type: Other; p = 0.060, Rao-Scott test

ADVERSE EVENTS:
Time Frame: Adverse event information was not applicable for this study.
Description: As this is a non-interventional study with secondary use of data from commercial and Medicare Advantage Part D (MAPD) beneficiaries, safety monitoring and safety reporting on an individual case level is not applicable. All-Cause Mortality, Serious Adverse Events and Other Adverse Events were not collected in the database. "0" total Number of Participants at Risk means "All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed".
Arm/Group | Tiotropium Bromide/Olodaterol (TIO/OLO) | Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/04/NCT05127304/Prot_SAP_000.pdf